CLINICAL TRIAL: NCT00503321
Title: Randomized Phase II Study of TS-1 Therapy and TS-1+PSK Therapy Against Unresectable Advanced Gastric Carcinoma and Recurrent Gastric Carcinoma
Brief Title: Phase II Study of TS-1 Therapy and TS-1+PSK Therapy Against Advanced Gastric Carcinoma
Acronym: eNCIT-Japan
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Patients' enrollment was not sufficient.
Sponsor: Eastern Network of Cancer Immunological Therapy, Japan (Other)
Responsible Party: Masanori Terashima, Shizuoka Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENCITJ-GC01
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer, TS-1, PSK
MeSH Terms: conditions — Stomach Neoplasms | interventions — Tegafur; S 1 (combination); polysaccharide-K

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B (Experimental): S-1 plus PSK group
  Interventions: Drug: Tegafur/gimeracil/oteracil potassium (S-1), Krestin (PSK)
- Arm A (Active Comparator): S-1 alone
  Interventions: Drug: Tegafur/gimeracil/oteracil potassium (S-1)

INTERVENTIONS:
Drug: Tegafur/gimeracil/oteracil potassium (S-1), Krestin (PSK) — S-1 80mg/m2 4weeks on 2 weeks off, PSK 3g/day
  Other Names: S-1 plus PSK
  Arms: Arm B
Drug: Tegafur/gimeracil/oteracil potassium (S-1) — S-1 80mg/m2, 4weeks on followed by 2 weks off
  Other Names: S-1 alone
  Arms: Arm A

SUMMARY:
A randomized controlled study is conducted on unresectable advanced gastric carcinoma and recurrent gastric carcinoma to compare TS-1 therapy with TS-1 + PSK therapy. The primary endpoint of this study is progression-free survival (PFS), with secondary endpoints of anticancer effect, time to treatment failure (TTF), QOL (FACT-BRM), compliance, adverse drug reactions and immunological factors.

DETAILED DESCRIPTION:
Tegafur / gimeracil / oteracil potassium (TS-1) is widely used as a first-line drug for unresectable advanced gastric carcinoma and recurrent gastric carcinoma in Japan and the response rate of TS-1 against gastric carcinoma was reported to be excellent at 46.5% in a phase II study. However, since adverse drug reactions tend to occur in patients treated with standard regimen of TS-1, drug reduction or discontinuation is often required, which is one drawback of this drug. On the other hand, although Krestin (PSK) has been reported to show survival effects in postoperative immunochemotherapy against gastric carcinoma, the efficacy of PSK has not been established in patients with unresectable advanced gastric carcinoma and recurrent gastric carcinoma. Since the main effect of PSK was to recover physiological functions, including immune function of the host, it was expected that PSK would improve the compliance of TS-1 by alleviating adverse drug reactions of TS-1 therapy and the concomitant use of TS-1 with PSK would result in the improvement of treatment results. Therefore, we decided to conduct a randomized phase II study on patients with unresectable advanced gastric carcinoma and recurrent gastric carcinoma to compare TS-1 therapy with TS-1+PSK therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable advanced gastric carcinoma and recurrent gastric carcinoma.
* Patients who are 20 years old or older at the time of obtaining consent.
* Patients who have not received prior treatment, including radiotherapy, chemotherapy and immunotherapy, before the start of treatment (however, patients are excluded when six months or more have passed since they received postoperative adjuvant chemotherapy.)
* Patients who do not develop metachronous or simultaneous multi cancer.
* Patients who do not show severe impairments in renal function, liver function and bone marrow function and who maintain the major organ functions which meet all requirements as described below (laboratory values are values measured before the start of protocol treatment and should be updated ones which are measured within two weeks before protocol treatment is started.) WBC counts: >= 3,000 /mm3 and < 12,000 /mm3 Neutrophil counts (ANC): >= 1,500 /mm3 Platelet counts: >= 100,000 /mm3 Amount of hemoglobin: >= 8.0 g/dL Serum GOT and GPT: Less than 100 IU/L Serum total bilirubin: Less than 1.5 mg/dL Serum creatinine: Less than 1.5 mg/dL
* Patients whose performance status scores are 0 to 2.
* Patients who are judged that they can endure this treatment in a comprehensive manner and who have provided written informed consent to participate in this research.
* Presence or absence of measurable lesion does not matter, but if there are measurable lesions in patients, the lesions should be confirmed within 28 days before the enrollment.

Exclusion Criteria:

* Patients with fresh blood in the digestive tract.
* Patients with body fluids which require treatment.
* Patients with infectious disease, intestinal paresis and ileus.
* Patients with diarrhea (watery stool).
* Female patients who are pregnant or want to become pregnant during this study or male patients who intend to make someone pregnant during this study.
* Diabetic patients who are being treated with insulin or are poorly controlled.
* Patients with ischemic heart disease which require treatment
* Patients who are complicated with psychosis and judged that it is difficult for them to participate in this study.
* Patients who continue to receive steroids.
* Patients who have experienced serious drug allergy in the past.
* Patients who are taking health foods including agaricus which are considered to have immunostimulating effects.
* Patients judged to be inappropriate for this study by investigators and sub-investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-10; Primary Completion 2009-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6 months

SECONDARY OUTCOMES:
Anticancer effect, time to treatment failure (TTF), QOL (FACT-BRM), compliance, adverse drug reactions and immunological factors | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hideaki Tahara, MD, Study Chair — Eastern Network of Cancer Immunological Therapy, Japan
Locations (1):
- Shizuoka Cancer Center, Shizuoka, Shizuoka, Japan

REFERENCES:
- [Background] Nakazato H, Koike A, Saji S, Ogawa N, Sakamoto J. Efficacy of immunochemotherapy as adjuvant treatment after curative resection of gastric cancer. Study Group of Immunochemotherapy with PSK for Gastric Cancer. Lancet. 1994 May 7;343(8906):1122-6. doi: 10.1016/s0140-6736(94)90233-x. PMID 7910230